CLINICAL TRIAL: NCT02189551
Title: Advanced Robotic Training With Additional Degrees of Freedom: Towards a Free-walking System
Acronym: LOKOMAT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: an additional intervention, amendet to the study (3rd arm, not described here), has not received clearance by regulatory authorities
Sponsor: Cereneo AG (Industry)
Collaborators: Swiss Commission for Technology and Innovation (Other); Swiss Federal Institute of Technology (Other); Hocoma AG (Unknown); University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: EKNZ: 2014-052
Record Dates: First submitted 2014-06-30; First posted 2014-07-14 (Estimated); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Post Stroke Gait Training

ARMS (2):
- Lokomat Pro (Active Comparator): gait robot established on the market
  Interventions: Behavioral: Gait training with Lokomat Pro
- Lokomat Pro FreeD (Experimental): gait robot based on the Lokomat Pro with changes in guidance of the hip, approved for the Swiss market
  Interventions: Behavioral: Gait training with Lokomat Pro FreeD

INTERVENTIONS:
Behavioral: Gait training with Lokomat Pro
  Arms: Lokomat Pro
Behavioral: Gait training with Lokomat Pro FreeD
  Arms: Lokomat Pro FreeD

SUMMARY:
The objective of the study is to compare a new medical devices with an established medical device for lower limb rehabilitation regarding training outcome and patient comfort / patient satisfaction (primary objective) and treatment effect (exploratory objective).

Primary study endpoints will be a significantly higher rated patient comfort and or patient satisfaction using the new versions, compared with the established Lokomat. Furthermore, muscle activity and kinematic movement patterns will be expected to show more involved muscle groups and a walking pattern involving more degrees of freedom during use of the new version compared with the established Lokomat.

Exploratory endpoints will be a significantly stronger involvement of muscles needed for balance, more physiological walking patterns and more change on the lateral positioning of the feet due to training with the new version, compared with the established Lokomat.

ELIGIBILITY:
Inclusion Criteria:

* Lower extremity weakness due to stroke
* minor functional impairment (MRC < 5)
* ability and willingness to participate

Exclusion Criteria:

* severe spasticity of the lower extremities
* severe dementia
* severe depression
* any other contraindications against Lokomat training
* body weight > 135 kg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2014-06; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Lateral hip movement | 30 min training during day 1 (next session after inclusion)
  during 30 min training with each device, lateral hip movements will be assessed

SECONDARY OUTCOMES:
Patient satisfaction | day 2 and 3
  Satisfaction, based on questionnaires, will be assessed after training with the experimental and the standard device in two consecutive sessions (randomized order).
Patient motivation | day 2 and 3
  Patient motivation, based on questionnaires, will be assessed after training with the experimental and the standard device in two consecutive sessions (randomized order).

CONTACTS AND LOCATIONS:
Locations (1):
- Cereneo, Center For Rehabilitation and Neurology, Vitznau, Canton of Lucerne, Switzerland